CLINICAL TRIAL: NCT05016856
Title: Adherence Promotion with Person-centered Technology (APPT): Promoting Adherence to Cognitive Intervention
Brief Title: Smart Reminders to Promote Home-based Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Walter Boot, Principal Investigator, Florida State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00000064
Record Dates: First submitted 2021-07-28; First posted 2021-08-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Adherence, Treatment
Keywords: adherence; cognitive intervention; memory support; artificial intelligence; aging; technology
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — 4-azido-7-phenylpyrazolo-(1,5a)-1,3,5-triazine; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Measures of adherence will be automatically collected and thus assessors will be blind to this outcome. Data will be coded and analyzed with arbitrary condition markers to mask condition during analysis. Participants will not be explicitly told which condition they are in, but will be aware of the reminder messages they are receiving, and thus are not truly blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reminder Only Condition (Active Comparator): To promote adherence, participants will receive generic reminders when home-based cognitive training has not been completed. This will be in the form of a text message to participants' smart phone.
  Interventions: Behavioral: Standard Reminder System (Active Control)
- Smart Adherence Support Condition (Experimental): To promote adherence, participants will receive reminders when home-based cognitive training has not been completed. This will be in the form of a text message to participants' smart phone. In this condition, participants will receive adaptive and tailored reminders based on dynamic algorithms that deploy reminders in a way that considers participant preferences, days and times of previous successful assessments, the success of previous reminder attempts, and answers to brief questions contained within reminder prompts. Parameter weights for these variables will be adjusted dynamically over a 6-month assessment period to ensure that reminders are deployed when they are most likely to be acted upon.
  Interventions: Behavioral: Adherence Promotion With Person-centered Technology (APPT) System

INTERVENTIONS:
Behavioral: Adherence Promotion With Person-centered Technology (APPT) System — A personalized and adaptive text message reminder system.
  Arms: Smart Adherence Support Condition
Behavioral: Standard Reminder System (Active Control) — A typical text message reminder system.
  Arms: Reminder Only Condition

SUMMARY:
This study will examine whether among older adults an adaptive and personalized reminder system can better support adherence to home-based cognitive training over typical reminder systems.

DETAILED DESCRIPTION:
Many cognitive training interventions are associated with poor adherence, and poor adherence is associated with fewer benefits. Further, poor adherence in cognitive intervention studies can interfere with answering fundamental questions regarding intervention efficacy. This study will compare the effects of non-adaptive and smart adherence support systems. Participants will be asked to engage in frequent home-based cognitive training on a computer tablet. In the smart adherence support condition, participants will receive adaptive and tailored reminders based on dynamic algorithms that deploy reminders in a way that considers participant preferences, days and times of previous successful engagement, the success of previous reminder attempts, and answers to brief questions contained within reminder prompts. Parameter weights for these variables will be adjusted dynamically over a 6-month assessment period to ensure that reminders are deployed when they are most likely to be acted upon. This study will investigate adherence to training sessions, multiple times each week for 6 months, representing a large challenge to adherence. Participants will be randomly assigned to one condition or another, and adherence at home will be monitored. This will be an Individually Randomized Group-Treatment Trial (IRGT).

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* normal or corrected to normal visual acuity
* must pass a dementia screening

Exclusion Criteria:

* Parkinson's, Alzheimer's disease, or any other neurodegenerative disease
* terminal illness
* blindness or deafness
* severe motor impairment
* not living in the Tallahassee area for the entire 6 month study period
* unable to read at or above 6th grade level

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 190 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Adherence (session number) | 6 months
  Number of sessions over 6 months
Adherence (session length) | 6 months
  Number of sessions reaching at least 80% of the assigned session duration over 6 months
Adherence (holidays) | 6 months
  Number of extended gaps in between sessions over 6 months

SECONDARY OUTCOMES:
Objective Cognition (predictor of adherence) | Assessed at baseline, predicting adherence variables over 6 months
  A composite measure of objective cognitive ability
Subjective Cognition (predictor of adherence) | Assessed at baseline, predicting adherence variables over 6 months
  A composite measure of subjective cognitive deficit
Self-Efficacy (predictor of adherence) | Assessed at baseline, predicting adherence variables over 6 months
  A composite measure of self-efficacy (beliefs held about ability to complete tasks)
Technology Proficiency (predictor of adherence) | Assessed at baseline, predicting adherence variables over 6 months
  A composite measure of proficiency with technology
Perceived Training Efficacy (predictor of adherence) | Assessed at baseline, predicting adherence variables over 6 months
  A composite measure of belief in the the efficacy of cognitive training
Personality (predictor of adherence) | Assessed at baseline, predicting adherence variables over 6 months
  Measure of stable traits
Dementia Worry (predictor of adherence) | Assessed at baseline, predicting adherence variables over 6 months
  A composite measure of anxiety over cognitive decline
Busyness Scale (predictor of adherence) | Assessed at baseline, predicting adherence variables over 6 months
  Self-reported environmental demands of day-to-day life

OTHER OUTCOMES:
Interview | 6 months
  Interview assessing experience in study

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified adherence data (time and date of intervention engagement) and scored individual difference measures (at the level of the individual) will be shared online.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available one year after the publication of the first primary outcome paper or two years after the collection of the final participants' data, whichever come first.
Access Criteria: Data will be freely available online.